CLINICAL TRIAL: NCT05077774
Title: Harmony TPV Post-Approval Study (Harmony PAS2)
Brief Title: Harmony TPV Post-Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20057CON003
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Tetrology of Fallot; RVOT Anomaly; Pulmonary Regurgitation
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Harmony TPV System (Other): Intervention Device: Harmony Transcatheter Pulmonary Valves and Delivery System
  Interventions: Device: Harmony TPV System

INTERVENTIONS:
Device: Harmony TPV System — Harmony Transcatheter Pulmonary Valve (sizes 22 mm and 25 mm) and Harmony Delivery Catheter System (DCS)
  Other Names: Model Numbers: HARMONY-22, HARMONY-25, and HARMONY-DCS

SUMMARY:
The purpose of this study is to characterize the functionality of transcatheter implantation of the Medtronic Harmony Transcatheter Pulmonary Valve (TPV) achieved by real-world implanters.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible to receive the Harmony TPV, meeting the indications for use criteria per current geography-specific device labeling at time of study enrollment
* Patient (or patient's legally authorized representative) is willing to consent to participate in the study

Exclusion Criteria:

* Obstruction of the central veins
* Planned concomitant branch pulmonary artery stenting at time of implant
* Subject is pregnant at time of implant procedure
* Patients with previously treated with an RV-PA conduit or previously implanted bioprosthesis
* A major or progressive non-cardiac disease (e.g. liver failure, renal failure, cancer) that results in a life expectancy of less than one year
* Planned implantation of the Harmony TPV in the left heart
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Pre-existing prosthetic heart valve or prosthetic ring in any position

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without valve reintervention and with acceptable hemodynamic function composite at 6 months as defined by: | 6 months
  * Mean RVOT gradient as measured by continuous-wave Doppler echocardiography ≤40 mmHg AND
  * Pulmonary regurgitant fraction as measured by CMR <20%

SECONDARY OUTCOMES:
Percentage of subjects free from all-cause mortality at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Percentage of subjects free from reoperation at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Percentage of subjects free from catheter reintervention at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Percentage of subjects free from TPV dysfunction at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Number and percentage of subjects with procedure success at 30-days | 30-days
Number and percentage of subjects with serious device-related adverse events at 6 months | 6 months
  Also described with Kaplan-Meier method for AEs of clinical interest.

CONTACTS AND LOCATIONS:
Overall Officials: David Balzer, MD, Principal Investigator — St. Louis Children's Hospital
Locations (20):
- United States (19):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - St. Joseph Children's Hospital, Tampa, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - The Mount Sinai Hospital, New York, New York
  - Children's Hospital New York - Presbyterian, New York, New York
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Children's Hospital, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Gillespie MJ, McElhinney DB, Jones TK, Levi DS, Asnes J, Gray RG, Cabalka AK, Fujimoto K, Qureshi AM, Justino H, Bergersen L, Benson LN, Haugan D, Boe BA, Cheatham JP. 1-Year Outcomes in a Pooled Cohort of Harmony Transcatheter Pulmonary Valve Clinical Trial Participants. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1917-1928. doi: 10.1016/j.jcin.2023.03.002. Epub 2023 May 17. PMID 37278682